CLINICAL TRIAL: NCT06379256
Title: Prospective Evaluation of Immune Responses and Outcomes in Patients With Hepatocellular Carcinoma Undergoing Radiotherapy
Brief Title: Evaluation of Immune Responses and Outcomes in Patients With Hepatocellular Carcinoma Undergoing Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202400364B0
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Photon Radiotherapy; Proton Radiotherapy; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Photons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Radiotherapy: Definitive photon or proton radiotherapy
  Interventions: Radiation: Photon or proton radiotherapy

INTERVENTIONS:
Radiation: Photon or proton radiotherapy — * 39.6-72.6 Gy (or Cobalt Gray Equivalent, CGE) in 22 fractions for tumors ≤1 cm from hepatic hilum, bowel, and heart.
  * 30-66 Gy (or CGE) in 10 fractions for tumors >1 cm from hepatic hilum, bowel, and heart.
  * 27.5-60 Gy (or CGE) in 5 fractions using stereotactic body radiation therapy (SBRT) techniques

SUMMARY:
Radiation therapy is a highly effective modality for managing localized solid tumors and has become a fundamental component of treating unresectable hepatocellular carcinoma. Our previous preclinical investigation revealed that radiotherapy can initiate immunogenic cell death and facilitate the cross-presentation of tumor antigens by antigen-presenting cells, thereby augmenting systemic anti-tumor T cell responses in murine tumor models. However, this immune response subsequent to irradiation has not been comprehensively evaluated in clinical trials involving hepatocellular carcinoma patients. Given that radiotherapy represents a standard therapeutic approach for unresectable hepatocellular carcinoma, our ongoing phase II non-randomized trial aims to prospectively assess immunological responses and dose-volumetric parameters, while identifying predictors of clinical outcomes in patients undergoing definitive radiotherapy for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have diagnosis of HCC. Participants may have multiple lesions. Diagnosis should be confirmed by at least 1 criteria listed below:

   * Histologically or cytologically proven diagnosis of HCC.
   * Typical arterial enhancement and delayed washout on multiphasic CT or MRI.
2. Age ≥18 years at the time of signing informed consent document.
3. ECOG performance status 0-2.
4. Child-Pugh score 5-9 liver function within 28 days of study registration.
5. Documented virology status of hepatitis B virus (HBV), as confirmed by screening HBV serology test.
6. Documented virology status of hepatitis C virus (HCV), as confirmed by screening HCV serology test.
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Presence of distant metastases that cannot be encompassed by radiotherapy
2. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
3. Inability to treat all sites of disease by radiotherapy
4. Known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine radiotherapy using photons or protons for HCC
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2029-03-17 (Estimated); Study Completion 2032-03-17 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 12 months
  PFS is defined as the time from signing the informed consent to the first occurrence of disease progression or death from any cause (whichever occurs first) according to RECIST1.1.

SECONDARY OUTCOMES:
Local control (LC) | 12 months
  LC is defined as the time from signing the informed consent to the first occurrence of disease progression in the irradiated field according to RECIST1.1.
Time to progression (TTP) | 12 months
  TTP is defined as the time from signing the informed consent to the first occurrence of disease progression according to RECIST1.1.
Overall Response Rate (ORR) | 12 months
  ORR is defined as a complete or partial response according to RECIST1.1.
Overall survival (OS) | 12 months
  OS is defined as the time from signing the informed consent to death from any cause.
Incidence and severity of adverse events | 12 months
  Adverse events will be graded using CTCAE v5

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data (IPD) with other researchers requires IRB review and approval. Presently, we do not have a plan to provide IPD to other researchers